CLINICAL TRIAL: NCT03206632
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 690517 in Healthy Chinese and Japanese Male Subjects (Double-blind, Randomised, Placebo-controlled Group Design)
Brief Title: This Study is Done in Healthy Chinese and Japanese Volunteers; it Looks at How BI 690517 is Taken up in the Body and How Well it is Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1378-0003
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BI 690517 dose group 1 (Experimental)
  Interventions: Drug: BI 690517
- BI 690517 dose group 2 (Experimental)
  Interventions: Drug: BI 690517
- BI 690517 dose group 3 (Experimental)
  Interventions: Drug: BI 690517
- Placebo (Placebo Comparator): Matching placebo for each dose group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 690517 — single dose
  Other Names: Vicadrostat
  Arms: BI 690517 dose group 1; BI 690517 dose group 2; BI 690517 dose group 3
Drug: Placebo — single dose
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 690517 in healthy Chinese and Japanese male subjects following oral administration of single doses.

Secondary objectives are the exploration of the pharmacokinetics (PK) including dose proportionality as well as the investigation of pharmacodynamic effects following single rising doses of BI 690517.

ELIGIBILITY:
Inclusion criteria

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Chinese ethnicity or Japanese ethnicity, according to the following criteria:

  * Chinese; born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in China
  * Japanese; born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who were all born in Japan
* Age of 20 to 45 years (incl.)
* Body Mass Index (BMI) of 18.5 to 25.0 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects who agree to minimize the risk of female partners being pregnant by fulfilling any of the following criteria starting from the first administration of trial medication and until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom: combined oral contraceptives, intrauterine device
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy) female partner

Exclusion criteria

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 60 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Values for serum sodium and potassium outside normal range at screening

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Number [N (%)] of subjects with adverse reactions | up to 336 hours

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 48 hours

OTHER OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea